CLINICAL TRIAL: NCT03816748
Title: The Efficacy of Postoperative Application of High Flow Nasal Cannula at Acute Phase for Minimally Invasive Esophagectomy Surgery Patients
Brief Title: The Efficacy of Postoperative Application of HFNC at Acute Phase for Minimally Invasive Esophagectomy Surgery Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201807098RINC
Record Dates: First submitted 2019-01-23; First posted 2019-01-25 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Esophageal Cancer
Keywords: Minimally invasive surgery; High flow nasal cannula
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention (Experimental): Patients who underwent minimally invasive esophagectomy surgery in our hospital and transfer to intensive care unit, and accept HFNC treatment
  Interventions: Device: High flow nasal cannula, HFNC
- control (No Intervention): Patients who underwent minimally invasive esophagectomy surgery in our hospital and transfer to intensive care unit, and accept usual care

INTERVENTIONS:
Device: High flow nasal cannula, HFNC — The HFNC used in this study can supply more than 40-60 L/min of oxygen flow, which is many times higher than the traditional nasal cannula. In addition, HFNC provides heating and moisturizing functions, so the patients 'nasal and oropharyngeal cavities do not dry out. This way, the patients can wear HFNC continuously for many days. Furthermore, when the patients close their mouths, HFNC can create a PEEP of 6-8 cmH2O, which helps with lung expansion after chest surgeries and lowers the risk of pneumonia related to lung collapses.
  Arms: intervention

SUMMARY:
This is a prospective study that uses the treatment guideline of our chest surgery ICU. Investigators recruited 90 patients who underwent MIE in the National Taiwan University Hospital. The clinical data collected included vital signs (blood pressure, heart rate, respiratory patterns and frequencies, saturation of blood oxygen and carbon dioxide, etc.), blood tests, images and bronchoscopic analysis of sputum.

The goal of this study is to analyze common care problems and complications patients may encounter during the acute stage in ICU after MIE. By comparing the differences between the treatment group and the control group, investigators can interpret the role of HFNC.

DETAILED DESCRIPTION:
In recent years, for resectable esophageal cancer lesions, the National Taiwan University Hospital has developed MIE from the traditional open-abdomen and open-chest reconstructive surgeries. Because the wounds of minimally invasive surgeries are smaller, most of the patients can be extubated soon in the operation rooms. During the period when the patients are sent to ICU for observation, they do not need endotracheal tubes for positive pressure or sputum suction. Thus, high standards are needed for the inspections of post-operative chest care, depth of respiration and ability of expectoration in these patients.

The HFNC used in this study can supply more than 40-60 L/min of oxygen flow, which is many times higher than the traditional nasal cannula. In addition, HFNC provides heating and moisturizing functions, so the patients 'nasal and oropharyngeal cavities do not dry out. This way, the patients can wear HFNC continuously for many days. Furthermore, when the patients close their mouths, HFNC can create a PEEP of 6-8 cmH2O, which helps with lung expansion after chest surgeries and lowers the risk of pneumonia related to lung collapses.

This is a prospective study that uses the treatment guideline of our chest surgery ICU. Investigators recruited 60 patients who underwent MIE in the National Taiwan University Hospital between January 2018 and December 2018. The clinical data collected included vital signs (blood pressure, heart rate, respiratory patterns and frequencies, saturation of blood oxygen and carbon dioxide, etc.), blood tests, images and bronchoscopic analysis of sputum.

The goal of this study is to analyze common care problems and complications patients may encounter during the acute stage in ICU after MIE. By comparing the differences between the treatment group and the control group, investigators can interpret the role of HFNC.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of esophageal cancer. Underwent minimally invasive esophagectomy surgery.

Exclusion Criteria:

1. The patient return to the intensive care unit without extubation 2. The patient who underwent tracheostomy surgery 3. Blood loss more than 1000c.c during the surgery 4. The patient who underwent CPR procedure or other emergent resuscitation management during surgery 5. The patient who is unable to communicate in words or speech

-

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Oxygenation | Post-operative 24 hours - 72 hours
  saturation of blood oxygen and carbon dioxide by blood gas analyzer

CONTACTS AND LOCATIONS:
Overall Officials: HSIEN-CHI LIAO, M.D., Study Director — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2017-08-07): https://cdn.clinicaltrials.gov/large-docs/48/NCT03816748/Prot_000.pdf